CLINICAL TRIAL: NCT03568058
Title: A Phase 1b Safety and Feasibility Study of Personalized Immunotherapy in Adults With Advanced Cancers
Brief Title: Personalized Immunotherapy in Adults With Advanced Cancers Immunotherapy in Adults With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ezra Cohen (Other)
Responsible Party: Sponsor-Investigator, Ezra Cohen, Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180410
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced Cancer
Keywords: immunotherapy; personalized cancer vaccine; personalized immunotherapy; pembrolizumab; Keytruda; cancer; neoantigen; solid tumor; vaccine
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- vaccine and anti-PD-1 (Experimental): personalized vaccine and anti-PD-1 administered concurrently at the start of study therapy
  Interventions: Drug: personalized vaccine; Drug: Pembrolizumab
- anti-PD1 before vaccine (Experimental): anti-PD-1 antibody for 6 weeks followed by personalized vaccine therapy
  Interventions: Drug: personalized vaccine; Drug: Pembrolizumab
- anti-PD1 and vaccine (Experimental): anti-PD-1 antibody followed by personalized vaccine therapy
  Interventions: Drug: personalized vaccine; Drug: Pembrolizumab
- vaccine (Experimental): personalized vaccine therapy
  Interventions: Drug: personalized vaccine

INTERVENTIONS:
Drug: personalized vaccine — Vaccine will be constructed for each subject that express multiple candidate tumor-derived neoantigens.
Drug: Pembrolizumab — 200 mg pembrolizumab will be administered intravenous (IV) infusion every 3 weeks.
  Other Names: keytruda
  Arms: anti-PD1 and vaccine; anti-PD1 before vaccine; vaccine and anti-PD-1

SUMMARY:
The purpose of this study is to determine if it is possible to make and administer safely a 'personalized' vaccine to treat patients that have been diagnosed with advanced cancer and are not candidates for curative therapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine if it is possible to make and administer safely a 'personalized' vaccine to treat patients that have been diagnosed with advanced cancer and are not candidates for curative therapy.

This 'personalized' vaccine will use information gained from specific characteristics of your own cancer. It is known that cancer has mutations (changes in genetic material) that are specific to an individual and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune (protective) responses, which may help your body fight any tumor cells that could cause your cancer to come back in the future. The study will examine the safety of the vaccine when given at several time points and will examine your blood cells for signs that the vaccine induced an immune response.

The personalized vaccine will be given in combination with an anti-PD1 antibody, pembrolizumab, which is used with the intention to increase anti-cancer immunity (protection). Pembrolizumab is a type of drug that blocks certain proteins made by some types of immune system cells, such as T cells, and some cancer cells. These proteins help keep immune responses in check and can keep T cells from killing cancer cells. When these proteins are blocked, the "brakes" on the immune system are released and T cells are able to kill cancer cells better.

This personalized vaccine is considered experimental because this is not an FDA approved therapy for cancer.

Pembrolizumab is FDA approved for the treatment of melanoma, non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), classical Hodgkin lymphoma (cHL), primary mediastinal large b-cell lymphoma (PMBCL), urothelial carcinoma, tumor mutational burden-high (TMB-H) cancer, cutaneous squamous cell carcinoma (cSCC), triple-negative breast cancer (TNBC), microsatellite instability-high (MSI-H) or mismatch repair deficient cancer, microsatellite instability-high or mismatch repair deficient colorectal cancer (CRC), gastric cancer, esophageal cancer, cervical cancer, and hepatocellular carcinoma (HCC), merkel cell carcinoma (MCC), renal cell carcinoma (RCC), endometrial carcinoma. Pembrolizumab is considered experimental (investigational) for the treatment of all other cancer types.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically documented incurable solid tumor [excluding lymphoma].
* Measurable disease as defined by RECIST 1.1
* Progressed on or be intolerant to therapies that are known to provide clinical benefit.
* Non-measurable disease by RECIST 1.1 and high-risk (>50% over 5 years) of mortality
* At least one tumor site accessible for biopsy.
* Adequate organ function
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria

* Currently receiving or has received another anti-cancer therapy within 4 weeks prior to first dose of vaccine study treatment.
* Currently receiving or has received PD1/PDL1 inhibitor immunotherapy within 4 weeks prior to first dose of study treatment.
* Currently receiving or has received anti-PD1 or anti-CTLA4 treatment during the vaccine preparation period.
* Receiving TNF pathway inhibitors, PI3 kinase inhibitors, systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study medication.
* Received an investigational agent within 28 days prior to the first dose of study drug.
* Untreated brain metastases; individuals with treated and stable metastases are eligible. Eligible subjects should have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for brain metastases for at least 4 weeks and are neurologically stable for 8 weeks (confirmed by MRI) prior to administration of experimental therapy
* Has known history of Human Immunodeficiency Virus (HIV).
* Received a diagnosis of hepatitis B or hepatitis C for which there is no clear evidence of natural immunity, immunity subsequent to vaccination, or successful eradication of the virus following antiviral therapy (individuals who are hepatitis C antibody positive may be enrolled if negative viral load confirmed).
* History of autoimmune disease including: inflammatory bowel disease (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g. Wegener's granulomatosis); central nervous system or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barré syndrome, myasthenia gravis, multiple sclerosis). Individuals with vitiligo, Sjogren's Syndrome, interstitial cystitis, Graves' or Hashimoto's Disease, celiac disease, DM1, or hypothyroidism stable on hormone replacement will be allowed with Study Medical Monitor's approval.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of receiving a solid organ transplant or allogeneic bone marrow transplant.
* Major surgical procedure within 28 days prior to the first dose of study drug.
* If female, pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative frequency of TCR | 1 year
  Quantitative frequency of TCR
Number of Participants with Treatment-related Adverse Events | 1 year
  Number of Participants with Treatment-related Adverse Events

SECONDARY OUTCOMES:
Overall Response | 1 year
  RECIST 1.1
Progression-free survival (PFS) | 1 year
  Duration of time from start of study treatment until objective tumor progression or death.
Time to Progression | 1 year
  Duration of time from start of study treatment until objective tumor progression.
Overall Survival | 1 year
  Duration of time from start of study treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Erza Cohen, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States